CLINICAL TRIAL: NCT03929718
Title: A Randomized Prospective Pilot Study to Evaluate Efficacy of Aldosterone Antagonist Therapy for Prevention of New Atrial Fibrillation (AF) in Patients With Atrial Flutter (AFL), But no Previously Detected AF, Undergoing caVOtricuspID Isthmus Ablation
Brief Title: Efficacy of Aldosterone Antagonist Therapy for Prevention of New Atrial Fibrillation
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVOID-AF
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: AFib
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: Randomized, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Therapy (Active Comparator): subjects undergoing CTI ablation
  Interventions: Drug: No Spironolactone
- Interventional Therapy (Experimental): subjects treated with an aldosterone antagonist after CTI ablation
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — receive spironolactone treatment after CTI ablation
  Arms: Interventional Therapy
Drug: No Spironolactone — no spironolactone treatment
  Arms: Standard Therapy

SUMMARY:
The purpose of this study is to accurately determine, using an implantable rhythm monitor, the long-term incidence of new atrial fibrillation after ablation of atrial flutter in those treated with spironolactone compared with standard medical therapy.

DETAILED DESCRIPTION:
Catheter ablation of the cavotricuspid isthmus (CTI) is an effective and safe procedure in patients with atrial flutter (AFL) with excellent long-term results in preventing AFL recurrences. However, new-onset atrial fibrillation (AF) commonly develops after this procedure and has important clinical implications for patient management. Few studies have assessed the long-term incidence and prevalence of AF after CTI ablation via intensive continuous rhythm monitoring with an implantable cardiac monitor. Furthermore, whether the development of AF can be impacted beneficially by adjunctive therapeutic approaches is not known. The co-primary objectives of this pilot study in patients with typical atrial flutter (AFL) but no previously detected AF are: 1) to accurately determine the long-term incidence of new-onset AF after CTI ablation using an implantable rhythm monitor; 2) to compare the rates of new onset AF in subjects randomized to standard, usual-care, medical therapy following CTI ablation compared with those randomized to treatment with an aldosterone antagonist (spironolactone) in addition to their usual care medications. The patient population will be subjects with typical atrial flutter and a history of hypertension or heart failure, but no known AF episodes, scheduled to undergo catheter ablation of the CTI for treatment of AFL. Patients will be randomized to remain on their standard, usual-care. medications or to take oral spironolactone (a standard, FDA-approved medication used in the treatment of hypertension and heart failure) starting after their ablation procedure. The primary study endpoint will be any atrial tachyarrhythmia episode (AF, AFL or atrial tachycardia) lasting greater than one minute detected via the implanted cardiac monitor after CTI ablation during long-term follow-up. The incidence of new-onset AF after CTI ablation will be compared between subjects randomized to be treated with usual care vs. those treated with usual care plus spironolactone on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of typical AFL confirmed by 12-lead ECG
* no documented AF on ECG, ambulatory monitor, pacemaker or ICD at any time
* scheduled to undergo catheter ablation of the CTI for treatment of AFL
* history of hypertension (HTN) or heart failure (HF) (reduced or preserved systolic function)

Exclusion Criteria:

* history of known AF episodes
* previous CTI or PVI ablation procedure
* other SVT mechanisms demonstrated (AVNRT, AVRT or accessory pathways)
* amiodarone usage within the past 3 months,
* unwillingness to participate or undergo insertable monitor implantation
* hyperkalemia (potassium > 5.0 mEq/L)
* severe renal disease (Cr >2.5 mg/dL [men], >2.0 mg/dL [women, GFR < 30 mL/min/1.73 m2)
* life expectancy < 18 months
* prior intolerance to treatment with an aldosterone antagonist
* current treatment with an aldosterone antagonist
* need for treatment with a class I or III AAD for another indication
* operative AFL (occurring within 30 days of surgery) that is expected to resolve
* presence of a cardiac rhythm device (pacemaker or ICD) capable of AF monitoring
* currently pregnant or nursing a child
* unwilling not to become pregnant and to use birth control while taking spironolactone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Long-Term incidence of new-onset AF after CTI ablation | 24 months
  1. To accurately determine the long-term incidence of new-onset AF after CTI ablation using an implantable rhythm monitor
Rates of new-onset AF between standard therapy and spironolactone | 24 months
  2. To compare the rates of new onset AF in subjects randomized to standard medical therapy following CTI ablation compared with those randomized to treatment with an aldosterone antagonist (spironolactone)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Stambler, MD, Principal Investigator — Piedmont Healthcare
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States